CLINICAL TRIAL: NCT00109174
Title: MRS (Magnetic Resonance Spectroscopy) Measurement of Glutamate and GABA Metabolism in Brain
Brief Title: MRS Measurement of Glutamate and GABA Metabolism in Brain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 050144; 05-M-0144
Record Dates: First submitted 2005-04-22; First posted 2005-04-25 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-08-08

CONDITIONS: Normal Physiology
Keywords: Glutamate; Excitatory Amino Acid; Neurochemistry; Brain; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- One arm (Other): Subjects receive the same test
  Interventions: Device: 3T and 7T device

INTERVENTIONS:
Device: 3T and 7T device — 3T and 7T device

SUMMARY:
This study will use magnetic resonance spectroscopy (MRS) to measure in the brain the transfer of [13]C as it is naturally metabolized from glucose to specific chemical transmitters. From this method, we can measure the rate of production of an important excitatory neurotransmitter (glutamate) as well as an inhibitory neurotransmitter (GABA)....

DETAILED DESCRIPTION:
13C is a stable (i.e., non-radioactive) isotope of carbon with a natural abundance of ~1%. Following infusion of [13C]glucose and/or [13C]acetate, in vivo MRS (magnetic resonance spectroscopy) can monitor the rate of flux of the 13C atom from glucose and/or acetate to glutamate to glutamine. Thus, this procedure can provide measure of glutamate (GLU) and glutamine (GLN) turnover in brain. We have established parameters to obtain these measurements in nonhuman primate brain. The current protocol seeks approval to optimize MRS parameters and to develop new MRS techniques for human brain using the GE 3T, the Siemens 3T, and the Siemens 7T device.

Study population: All subjects will be aged 18 65 years, without serious medical illnesses and meet criteria listed in Section VI A.

Design: Subjects will receive either oral administration of [13C]glucose or an intravenous infusion of [13C]glucose and/or [13C]acetate to approximately double their plasma glucose levels. The plasma acetate level will remain within the physiological range observed in humans (Lebon et al, 2002). While lying in the 3T or 7T device, serial data acquisitions will be obtained over ~2 h to optimize the experimental conditions so as to measure the 13C signals from GLU, GLN and other metabolisms in brain.

Outcome measures: The primary goal of this study is to measure GLU/GLN turnover in brain. With no additional data acquisition, we can also obtain information on the synthesis of GABA, the major inhibitory neurotransmitter in brain. GLU is converted to GABA via the enzyme glutamic acid decarboxylase (GAD). While monitoring the transfer of 13C signal from GLU to GLN, we can simultaneously measure the transfer of 13C signal from GLU to GABA and thereby measure the activity of GAD (Li et al 2005). In addition to directly measure 13C signals, 13C labeling to brain metabolites can also be measured indirectly by detecting proton MRS during infusion of [13C]glucose and/or [13C]acetate.

ELIGIBILITY:
* INCLUSION CRITERIA:
* 18-65 years of age
* Able to give written informed consent
* Healthy based on medical history and physical exam
* Enrolled in Protocol 01-M-0254 or Protocol 17-M-0181

EXCLUSION CRITERIA:

* Any current Axis 1 diagnosis
* Clinically significant laboratory abnormalities
* Positive HIV test
* Metallic foreign bodies that would be affected by the magnetic resonance imaging (MRI) magnet, or fear of enclosed spaces likely to make the subject unable to undergo an MRI scan.
* History of neurological illness or injury with the potential to affect study data interpretation, such as multiple sclerosis, Parkinson s disease, seizure disorder or traumatic brain injury
* Prescription psychotropic medication; drug free less than 8 weeks (anticholinergics, benzodiazepine, fluoxetine, antipsychotics, and anticonvulsants)
* Serious medical illness as determined from H&P or laboratory testing including Diabetes
* Inability to lie flat on camera bed for about two and a half hours
* Pregnant or breastfeeding
* Current substance use disorder based on DSM-5
* NIMH employees and staff and their immediate family members will be excluded from the study per NIMH policy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-09-06 (Actual); Primary Completion 2030-01-11 (Estimated); Study Completion 2030-03-11 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the quality of the MR spectroscopy which includes spectrum signal-to-noise (SNR)\ ratio, spectral lineshape, linewidth, and resolution. | prospective and ongoing
  To obtain more accurate and reliable MRS data from the human brain

SECONDARY OUTCOMES:
The secondary outcome is the performance improvements of the scanner hardware, software and methodology | prospective and ongoing
  To obtain more accurate and reliable MRS data from the human brain.

CONTACTS AND LOCATIONS:
Overall Officials: Li An, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2005-M-0144.html